CLINICAL TRIAL: NCT02407860
Title: Efficacy of an Osteopathic Treatment for Mechanical Sucking Dysfunctions in Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Isabelle Gaboury, Assistant professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-116
Record Dates: First submitted 2015-03-10; First posted 2015-04-03 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Breastfeeding
Keywords: breast feeding; sucking; dysfunction; Latch assessment tool; visual analogic scale; infant physiology
MeSH Terms: conditions — Breast Feeding | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment (Experimental): one single osteopathic treatment in addition to usual breastfeeding counselling
  Interventions: Other: osteopathic treatment
- control (Active Comparator): usual breastfeeding counselling. Osteopathic evaluation of entire body
  Interventions: Other: usual breastfeeding counselling

INTERVENTIONS:
Other: osteopathic treatment — Treatment duration range between 30 to 40 minutes. The infant entire body is evaluated and then manipulative procedures are provided following palpatory results.
  Arms: treatment
Other: usual breastfeeding counselling — breastfeeding counselling and support by lactation consultant
  Arms: control

SUMMARY:
Breastfeeding is the physiological and recommended way of feeding newborns as indicated by the World Health Organization, Health Canada and the politics of perinatality 2008-2018 in Quebec. Despite these, mothers who exclusively breastfed their babies are rare. According to Statistics Canada, the first month of life is the most at risk time to wean because of technical difficulties (53% of weaning) including mechanical issues. In Quebec city, despite a supportive network of health care professionals including lactation consultant, many babies are weaned. Lactation consultant are often feeling helpless when facing these mechanical difficulties.

The purpose of this study is to determine the efficiency of an osteopathic treatment for newborns presenting breastfeeding mechanical difficulties. The investigators' hypotheses is that an osteopathic treatment integrating in the usual care is more efficient than usual car alone to help healing mechanical breastfeeding issues.

The investigators propose a randomized clinical trial on a sample of 90 babies (45 in each group), under six weeks, presenting sucking dysfunctions, in Quebec city (Canada). The control group will receive usual care with a lactation consultant and the intervention group will receive usual care plus an osteopathic treatment. It is a simple blind clinical trial: the osteopath finds out, prior to evaluating the patient, what intervention should be delivered to the baby (assessment alone or standardized osteopathic treatment for infant).

The results will ultimately lead to improvements in the existing knowledge on the fields of osteopathy and lactation support, allowing implementation of osteopathic care in the perinatal network.

ELIGIBILITY:
Inclusion Criteria:

* healthy term newborn,
* mechanical suckling dysfunction, assessed by lactation consultant or midwives or healthcare professionals with breastfeeding experience.

Exclusion Criteria:

* breastfeeding difficulties from mother (hypogalactia, breast hypoplasia, medication),
* twins or more,
* tongue-tie or lip tie pending for surgical treatment,
* previous or current bodywork (chiropractic, osteopathy, physiotherapy, ergotherapy, craniosacral therapy).

Ages: 48 Hours to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in baby's latch at the breast | Immediately after the intervention and 2 days post-intervention
  Latch assessment tool (Jensen, Wallace & Kelsay; 1994)

SECONDARY OUTCOMES:
Change from baseline in numbers of feeds per day | Immediately after the intervention and 2, and 10 days post-intervention
  Home made questionnaire with close-ended questions
Change from baseline in devices used to feed the baby | 2 and 10 days post-intervention
  Home made questionnaire with open-ended and close-ended questions, including the number of bottles the day before.
Change from baseline in mother's nipple pain | Immediately after the intervention and 2, and 10 days post-intervention
  Visual analog scale from 0 (no pain) to 10 (extreme pain)
Change from baseline in baby's head rotation | Immediately after the intervention
  Assessment of baby's ability to rotate his/her head on left and right compared to a baseline evaluation prior to the intervention, using a goniometer
Mother's satisfaction with an osteopathic approach | 10 days post-intervention
  Likert scale to assess the mother's perception of an osteopathic approach with four items: not at all satisfied, somewhat satisfied, satisfied and very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Gaboury, PhD, Study Director — Université de Sherbrooke
Locations (1):
- Entraide Naturo-Lait, Québec, Quebec, Canada